CLINICAL TRIAL: NCT01131299
Title: Evaluation of Oral Alpha-Cyclodextrin for Decreasing Serum Cholesterol
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Marcelo Amar, M.D., Medical Officer (Research), National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 100088; 10-H-0088 (Other: NIH NHLBI)
Record Dates: First submitted 2010-05-25; First posted 2010-05-26 (Estimated); Results first posted 2016-10-21 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-10

CONDITIONS: Cardiovascular Disease
Keywords: HDL; Cholesterol; Lipoproteins; Serum Lipids; Alpha-Cyclodextrin; Atherosclerosis; Heart Disease
MeSH Terms: conditions — Cardiovascular Diseases; Atherosclerosis; Heart Diseases | interventions — alpha-cyclodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Alpha cyclodextrin first then placebo (Active Comparator): Randomized subjects will receive alpha cyclodextrin 2g orally three times a day for 12-14 weeks. After the one week washout, the subjects will receive 2 tablets orally of placebo (three times a day for 12-14 weeks).
  Interventions: Other: Placebo; Drug: Alpha cyclodextrin
- Placebo first then Alpha cyclodextrin (Placebo Comparator): Participants will receive 2 tablets orally of placebo (three times a day for 12-14 weeks). The subjects will have a one-week washout. After the washout, the participants will receive alpha cyclodextrin 2g orally three times a day for 12-14 weeks.
  Interventions: Other: Placebo; Drug: Alpha cyclodextrin

INTERVENTIONS:
Other: Placebo — 2 tablets PO 3 times a day for 12-14 weeks
Drug: Alpha cyclodextrin — 2g PO 3 times a day for 12-14 weeks
  Other Names: alpha- CD; Alpha-CD

SUMMARY:
Background:

* Cardiovascular disease (CVD) is a leading cause of death in developed countries. Although statin-type drugs are currently the most effective therapeutic agents for reducing CVD risk. One possible complementary approach involves the use of soluble dietary fibers that are known to reduce blood cholesterol levels. However, analysis has shown that most soluble fibers reduce total cholesterol levels by relatively small amounts.
* Alpha-Cyclodextrin (Alpha-CD), also sold in commerical form, is a soluble fiber derived from corn that is used as an ingredient in many foods, such as bread rolls, crackers, juices, and reduced fat spreads. It is added to food primarily as a fiber supplement but is also used to stabilize flavors, colors, vitamins, and fatty acids. Studies in animals and humans have shown that Alpha-CD may help to improve insulin resistance and lower LDL cholesterol levels with no apparent side effects. More research is needed to determine the effect of Alpha-CD on total cholesterol levels in healthy volunteers.

Objectives:

- To determine the effect of oral Alpha-CD on total cholesterol in a nondiabetic population.

DETAILED DESCRIPTION:
This single center, double-blinded, cross-over, placebo controlled clinical pilot study will investigate the effectiveness of a soluble dietary fiber, alpha-cyclodextrin (alpha-CD), on blood lipid and lipoprotein levels in healthy human subjects. alpha-CD, a cyclical polymer of glucose, is currently sold as an over the counter food supplement and is a common ingredient in many foods. This is the first study that will evaluate the effect of alpha-CD in healthy subjects. One gram of alpha-CD has been shown to bind as much as 9 grams of dietary fat, and like other soluble dietary fibers or bile acid sequestrants (BAS) it may decrease the intestinal absorption of fats, which has been shown to reduce the incidence of cardiovascular disease (CVD). Animal studies in our laboratory have shown that oral alpha-CD lowers Low Density Lipoprotein-cholesterol (LDL-C) by approximately 15 percent in mice on a high fat diet. Other clinical trials utilizing this compound showed that it is a safe therapy with no significant side effects.

Eligibility:

- Individuals between 18 and 75 years of age who do not have type 1 or type 2 diabetes.

Design:

* This study will require three visits to the NIH Clinical Center.
* At the first visit, participants will provide information about current diet and exercise routines, and will have a physical examination with blood and urine tests. At the end of this visit, participants will be randomized to receive either Alpha-CD or placebo, and will be asked to take two 1 gram tablets three times a day, anytime from 1 hour before to the end of each meal. Participants will take a total of six tablets per day for 12 weeks.
* At the end of the first 12 weeks, participants will return to the clinical center for another interview and examination, and blood and urine tests. At the end of this visit, participants will receive the treatment not given in the first part of the study (either Alpha-CD or placebo), and will take tablets on the same schedule as before for 12 more weeks.
* Participants will wait for 1 week after stopping the previous study prescription before starting the next one.
* At the end of the second 12 weeks, participants will have a final interview and examination with blood and urine tests.
* Participants will be asked to keep 7-day food records before each clinic visit to be collected at the second and third visits. A short physical activity assessment will be collected at each visit to review any changes in physical activity.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Males and females between the ages of 18-75.

Subject understands protocol and provides written, informed consent in addition to a willingness to comply with specified follow-up evaluations.

EXCLUSION CRITERIA:

* Pregnancy or women currently breastfeeding.
* BMI less than 18.5
* Subjects with unstable weight that varies greater than 10% over the past 3 months.
* Subjects currently following any low-fat (< 20%) diet.
* Subjects that routinely consume less than 3 meals/snacks per day
* Subjects taking the following medications, which may show reduced absorption with alpha-CD or may otherwise interfere with the study will be excluded: soluble fiber supplements, BAS, plant sterol supplements, antibiotics, anticoagulants, anticonvulsants, antiarrhythmics , cyclosporine, mycophenolate, synthroid, vitamin A, E and K and or any drug that is necessary to take with a meal. If any of these medications are initiated during the study, the subjects will be instructed to discontinue the use of the alpha-CD or placebo pills and to withdraw from the study. Short-term and prophylactic antibiotics may be taken during study participation for up to 14 days, at least 2 hours apart from the study drug.
* Subjects with chronic diarrhea, gastric bypass or lap-band procedures, ostomies, bowel motility problems, or other conditions that could affect intestinal fat absorption.
* Subjects initiating new medications or patients on multiple medications may also be excluded.
* Patients with type I or type II diabetes.
* Subjects currently taking alpha-CD in its commercial form.
* Volunteers may also be excluded, if in the opinion of the study investigators, they have some other condition or disorder that may adversely affect the outcome of the study or the safety of the volunteer.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2010-03; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo J Amar, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fedder DO, Koro CE, L'Italien GJ. New National Cholesterol Education Program III guidelines for primary prevention lipid-lowering drug therapy: projected impact on the size, sex, and age distribution of the treatment-eligible population. Circulation. 2002 Jan 15;105(2):152-6. doi: 10.1161/hc0202.101971. PMID 11790693
- [Background] Cannon CP, Braunwald E, McCabe CH, Rader DJ, Rouleau JL, Belder R, Joyal SV, Hill KA, Pfeffer MA, Skene AM; Pravastatin or Atorvastatin Evaluation and Infection Therapy-Thrombolysis in Myocardial Infarction 22 Investigators. Intensive versus moderate lipid lowering with statins after acute coronary syndromes. N Engl J Med. 2004 Apr 8;350(15):1495-504. doi: 10.1056/NEJMoa040583. Epub 2004 Mar 8. PMID 15007110
- [Background] Shepherd J. Dyslipidaemia in diabetic patients: time for a rethink. Diabetes Obes Metab. 2007 Sep;9(5):609-16. doi: 10.1111/j.1463-1326.2006.00642.x. PMID 17697054
- [Derived] Amar MJ, Kaler M, Courville AB, Shamburek R, Sampson M, Remaley AT. Randomized double blind clinical trial on the effect of oral alpha-cyclodextrin on serum lipids. Lipids Health Dis. 2016 Jul 12;15(1):115. doi: 10.1186/s12944-016-0284-6. PMID 27405337
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2010-H-0088.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment occurred at the Clinical Center, NIH.
Pre-assignment Details: 103 screened participants, 75 completed the study, 14 subject withdrawals and 14 subjects who did not meet inclusion criteria
Groups:
- Placebo First, Then Alpha Cyclodextrin: Randomized subjects will receive placebo 2 tablets orally (three times a day) for 12-14 weeks. After a one-week washout, the subjects will receive alpha cyclodextrin.
  Alpha cyclodextrin: 2 tablets PO 3 times a day for 12-14 weeks
- Alpha Cyclodextrin First, Then Placebo: Subjects will receive alpha cyclodextrin: 2 tablets PO 3 times a day for 12-14 weeks. After a one-week washout, the subjects will receive placebo.
  Subjects will receive placebo 2 tablets orally (three times a day) for 12-14 weeks
Period: Overall Study
Arm/Group | Placebo First, Then Alpha Cyclodextrin | Alpha Cyclodextrin First, Then Placebo
Started | 42 | 44
Completed | 38 | 37
Not Completed | 4 | 7
Not completed — Withdrawal by Subject | 4 | 7

BASELINE CHARACTERISTICS:
Groups:
- Alpha Cyclodextrin & Placebo Participants: Randomized subjects receiving alpha cyclodextrin
  Alpha cyclodextrin: 2 g PO 3 times a day for 12- 14 weeks
  Randomized subjects receiving placebo comparator
  Placebo: 2 tablets PO 3 times a day for 12-14 weeks
Arm/Group | Alpha Cyclodextrin & Placebo Participants
Number analyzed (Participants) | 103
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 99
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60
  Male | 43
Region of Enrollment [Number; unit: participants]
  United States | 103

OUTCOME MEASURES:

1. Primary Outcome: Total Serum Cholesterol Levels for Alpha-cyclodextrin (a-CD) and Placebo Groups After 12-14 Weeks, Compared to Baseline
Description: Total cholesterol levels were measured at the end of each study arm (a-CD or placebo). a-CD (2g) was taken orally three times a day for 12-14 weeks. Placebo (2 tablets) was taken orally for 12-14 weeks. There was a one-week washout period between each arm.
Time Frame: 24-28 weeks
Measure: Mean (Standard Error); unit: mg/dL
Groups:
- a-CD; Placebo: Change in total serum cholesterol after 12-14 weeks intervention, compared to baseline
Arm/Group | a-CD | Placebo
Number analyzed (Participants) | 75 | 75
mg/dL | 180 (4) | 180 (4)
Statistical Analysis 1: Comparison: a-CD vs Placebo; The minimum sample size to detect an 8 mg/dl change in total plasma cholesterol between the placebo and alpha cyclodextrin periods is 62 subjects. The power is 80% by using the normal approximation to a one-sample (paired) two-tail t-test at an alpha of 0.05; Test type: Superiority or Other; p = 0.82, t-test, 2 sided

2. Secondary Outcome: Small LDL Particle Number (by NMR Spectrometry of Lipoproteins) After 12-14 Weeks Intervention, Compared to Baseline for Alpha-cyclodextrin (a-CD) and Placebo Groups After 12-14 Weeks, Compared to Baseline
Description: Small LDL particle numbers were measured at the end of each study arm (a-CD or placebo). a-CD (2g) was taken orally three times a day for 12-14 weeks. Placebo (2 tablets) was taken orally for 12-14 weeks. There was a one-week washout period between each arm.
Time Frame: 24-28 weeks
Measure: Mean (Standard Error); unit: nmol/L
Arm/Group | a-CD | Placebo
Number analyzed (Participants) | 75 | 75
nmol/L | 365 (35) | 405 (38)
Statistical Analysis 1: Comparison: a-CD vs Placebo; Test type: Superiority or Other; p = 0.04, t-test, 2 sided

3. Secondary Outcome: Serum Glucose Levels After 12-14 Weeks Intervention, Compared to Baseline for Alpha-cyclodextrin (a-CD) and Placebo Groups After 12-14 Weeks, Compared to Baseline
Description: Serum glucose levels was measured at the end of each study arm (a-CD or placebo). a-CD (2g) was taken orally three times a day for 12-14 weeks. Placebo (2 tablets) was taken orally for 12-14 weeks. There was a one-week washout period between each arm.
Time Frame: 24-28 weeks
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | a-CD | Placebo
Number analyzed (Participants) | 75 | 75
mg/dL | 87 (0.7) | 88 (0.9)
Statistical Analysis 1: Comparison: a-CD vs Placebo; Test type: Superiority or Other; p = 0.05, t-test, 2 sided

4. Secondary Outcome: Lipoprotein Insulin Resistance Index (LIRI) After 12-14 Weeks Intervention, Compared to Baseline for Alpha-cyclodextrin (a-CD) and Placebo Groups After 12-14 Weeks, Compared to Baseline
Description: LIRI was measured at the end of each study arm (a-CD or placebo). a-CD (2g) was taken orally three times a day for 12-14 weeks. Placebo (2 tablets) was taken orally for 12-14 weeks. There was a one-week washout period between each arm.
Time Frame: 24-28 weeks
Population: The LIRI score is a composite of six lipoprotein parameters (VLDL, HDL and LDL, and concentrations of large VLDL, large HDL and small LDL subclasses) measured by NMR spectroscopy, which may be apparent years before the onset of overt hyperglycemia. LIRI scores range from zero, the most insulin sensitive, to 100, the most insulin resistant.
Measure: Mean (Standard Error); unit: percentage
Arm/Group | a-CD | Placebo
Number analyzed (Participants) | 75 | 75
percentage | 1.4 (0.1) | 1.6 (0.1)
Statistical Analysis 1: Comparison: a-CD vs Placebo; Test type: Superiority or Other; p = 0.04, t-test, 2 sided

ADVERSE EVENTS:
Groups:
- Entire Study Population: Randomized subjects receiving active comparator
  Alpha cyclodextrin: 2g PO 3 times a day for 12-14 weeks
  Randomized subjects receiving placebo comparator
  Placebo: 2 tablets PO 3 times a day for 12-14 weeks
Arm/Group | Entire Study Population
Serious Adverse Events (participants affected / at risk) | 2/75
Other Adverse Events (participants affected / at risk) | 14/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Entire Study Population (N=75)
appendectomy (Gastrointestinal disorders) | 1
enrollment in conflicting clinical trial (Social circumstances) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1.33% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Entire Study Population (N=75)
abdominal pain (Gastrointestinal disorders) | 2 (2)
intestinal gas (Gastrointestinal disorders) | 3 (3)
nausea (Gastrointestinal disorders) | 1 (1)
diarrhea (Gastrointestinal disorders) | 3 (3)
urinary urgency (Renal and urinary disorders) | 1 (1)
dyspepsia (indigestion) (Gastrointestinal disorders) | 2 (2)
abdominal cramps (Gastrointestinal disorders) | 1 (1)
urinary frequency (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes